CLINICAL TRIAL: NCT06611189
Title: A Comparative Analysis of Ray-Tech Sponge and Ice Bag Techniques in the Elimination of Warm Ischemic Time in Kidney Transplantation
Brief Title: A Comparative Analysis of Ray-Tech Sponge and Ice Bag Techniques in Kidney Transplantation
Status: Active, not recruiting | Type: Observational
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Murat Ferhat Ferhatoglu, Principal Investigator, Okan University
Other Study IDs: No: 161, Date: December 14, 20
Record Dates: First submitted 2024-09-10; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Chronic Kidney Disease Stage V
Keywords: Kidney transplantation; Warm ischemia
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Kidney transplantation performed using the ice bag technique.
  Interventions: Other: surgery
- Group B: Kidney transplantation performed using Raytech sponge technique.
  Interventions: Other: Ray-Tech sponge technique

INTERVENTIONS:
Other: surgery — In order to preserve kidney from warm ischemia during graft implantation, on the back table, graft were prepared for implantation with standard techniques. The kidney was introduced into the bag which was filled with a small amount of ice and preservation fluid (Figure 1). After inplacement of the graft, a small hole was made near the hilum and the renal artery and vein were passed through the hole. A Kocher clamp was used to maintain the fluid and ice in place and as a handle. Also, a Hartman Mosquito Clamp was used to mark urether-side, and to maintain orientation.
  Other Names: Simple plastic bag to preserve kidney from warm ischemia
  Groups: Group A
Other: Ray-Tech sponge technique — On the back table, graft were prepared for implantation with standard techniques. A Raytech sponge is soaked in ice-cold preservative solution, and wrapped around the kidney and held with a clamp (Figure 2). Position and oriantation of the graft was done by direct vision of urether.
  Groups: Group B

SUMMARY:
Warm ischemia during kidney transplantation is one of the important factors that negatively affect kidney function in the recipient. The investigators aimed to examine the effects of two techniques (Ray-Tech sponge technique and Ice bag technique) applied to protect the kidney from warm ischemia during kidney transplantation on long-term kidney function.

DETAILED DESCRIPTION:
A prospective, randomized clinical trial was conducted at Istanbul Okan University Hospital, Istanbul, Turkey. All participants were selected from those who underwent kidney transplantation between January 2020 and January 2023.

ELIGIBILITY:
Inclusion Criteria:

-Underwent kidney transplantation surgery

Exclusion Criteria:

- Deceased donor transplantation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All individuals were selected from those who underwent Kidney transplantation at our institution between January 2020 and January 2023.
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Creatinine decrease | 6 months
  Serum creatinine levels at 7th, 30th, 60th, and 180th days after operation were evaluated

CONTACTS AND LOCATIONS:
Overall Officials: MURAT F FERHATOGLU, MD, Principal Investigator — Okan University
Locations (2):
- Turkey (Türkiye) (2):
  - Murat Ferhat Ferhatoglu, Istanbul, Kadıköy
  - Istanbul Okan University, Istanbul

IPD SHARING:
Plan to Share IPD: No
Sharing data is not right in terms of patient privacy. When the informed consent form was signed by participants, only information about the study was given. No information was given about data sharing.

REFERENCES:
- [Background] Ferede AA, Walsh AL, Davis NF, Smyth G, Mohan P, Power R, Forde J, O'Kelly P, Llittle D. Warm Ischemia Time at Vascular Anastomosis is an Independent Predictor for Delayed Graft Function in Kidney Transplant Recipients. Exp Clin Transplant. 2020 Feb;18(1):13-18. doi: 10.6002/ect.2018.0377. Epub 2019 Jul 2. PMID 31266437
- [Background] Ide K, Sakai H, Nakano R, Imaoka Y, Tanimine N, Ide R, Tsukiyama N, Ono K, Mochizuki T, Arata R, Hakoda K, Imaoka K, Fukuhara S, Bekki T, Tahara H, Ohira M, Kobayashi E, Ohdan H. Effectiveness of Thermal Barrier Bag for Prolonged Vascular Anastomosis in Kidney Transplantation. Transplant Proc. 2023 May;55(4):752-755. doi: 10.1016/j.transproceed.2023.03.004. Epub 2023 Apr 6. PMID 37028949
- [Background] Ide K, Nakano R, Imaoka Y, Sakai H, Ono K, Tanimine N, Tahara H, Ohira M, Ueda K, Hirata T, Kobayashi E, Ohdan H. Protection From Second Warm Ischemic Injury Using a Thermal Barrier Bag in Kidney Transplantation. Transplant Direct. 2023 Feb 17;9(3):e1454. doi: 10.1097/TXD.0000000000001454. eCollection 2023 Mar. PMID 36845857